CLINICAL TRIAL: NCT02286921
Title: A Randomized Phase II Study Comparing Bipolar Androgen Therapy vs. Enzalutamide in Asymptomatic Men With Castration Resistant Metastatic Prostate Cancer
Brief Title: Testosterone Revival Abolishes Negative Symptoms, Fosters Objective Response and Modulates Enzalutamide Resistance
Acronym: Transformer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J14146; IRB00046414 (Other: JHU IRB); W81XWH-14-2-0189 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2014-10-22; First posted 2014-11-10 (Estimated); Results first posted 2019-05-01 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-07

CONDITIONS: Castration Resistant Metastatic Prostate Cancer
Keywords: Testosterone; Enzalutamide; Abiraterone; Androgen Ablative Therapies; Bipolar Androgen Therapy
MeSH Terms: interventions — testosterone 17 beta-cypionate; enzalutamide; testosterone enanthate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Testosterone cypionate or testosterone enanthate (Experimental): Patients on BAT will receive testosterone cypionate or testosterone enanthate administered as an intramuscular injection. A dose of 400 mg of either agent will be injected intramuscularly (IM) every 28 days.
  Interventions: Drug: Testosterone cypionate; Drug: Testosterone Enanthate
- Arm B: Enzalutamide (Experimental): Patients randomized to enzalutamide will be prescribed enzalutamide 40 mg tablets and instructed to take 4 tablets per day orally for 28 days/cycle.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Testosterone cypionate — Depo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble of the androgenic hormone testosterone. Testosterone cypionate is a white or creamy white crystalline powder, odorless or nearly so and stable in air. Depo-Testosterone Injection is available in two strengths, 100 mg/mL and 200 mg/mL testosterone cypionate.
  Other Names: Depo-Testosterone Injection
  Arms: Arm A: Testosterone cypionate or testosterone enanthate
Drug: Enzalutamide — Enzalutamide is a white crystalline non-hygroscopic solid. It is practically insoluble in water. Enzalutamide is provided as liquid-filled soft gelatin capsules for oral administration. Each capsule contains 40 mg of enzalutamide as a solution in caprylocaproyl polyoxylglycerides. The inactive ingredients are caprylocaproyl polyoxylglycerides, butylated hydroxyanisole, butylated hydroxytoluene, gelatin, sorbitol sorbitan solution, glycerin, purified water, titanium dioxide, and black iron oxide.
  Other Names: Xtandi
  Arms: Arm B: Enzalutamide
Drug: Testosterone Enanthate — Testosterone Enanthate Injection, for intramuscular injection, contains testosterone enanthate which is the oil-soluble ester of the androgenic hormone testosterone. Enanthate Injection is available as a colorless to pale yellow solution. Each mL contains 200 mg testosterone enanthate in sesame oil with 5 mg chlorobutanol as a preservative.
  Other Names: Delatestryl
  Arms: Arm A: Testosterone cypionate or testosterone enanthate

SUMMARY:
Asymptomatic men with progressive metastatic Castration-resistant prostate cancer (CRPC) post- treatment with abiraterone acetate (pre-chemotherapy for metastatic disease) will be treated on a randomized, multi-Institutional open label study to determine if treatment with intramuscular T given on a dose/schedule designed to result in rapid cycling from the polar extremes of supraphysiologic to near castrate levels [i.e. Bipolar Androgen Therapy (BAT)] will improve primary and secondary objectives vs. enzalutamide as standard therapy.

DETAILED DESCRIPTION:
Eligible patients will have metastatic CRPC with no disease related symptoms and progression on Androgen deprivation therapy and will have progressed post-treatment with abiraterone. Patients will continue on Androgen deprivation therapy with Luteinising Hormone Releasing Hormone agonist (i.e. Zoladex, Trelstar, Eligard or Lupron) or Luteinising Hormone Releasing Hormone antagonist (Degarelix) if not surgically castrated throughout the duration of the study to inhibit endogenous testosterone production. Patients will be randomized 1:1 and stratified based on duration of prior abiraterone acetate therapy (6 months or less or greater than 6 months). Patients randomized to BAT (Arm A) will receive intramuscular injections with either testosterone cypionate or testosterone enanthate at a dose of 400 mg every 28 days. This dose was selected based on data demonstrating that it produces an initial supraphysiologic serum level of T (i.e. > 1500 ng/dL or 3-10 times normal level) with eugonadal levels achieved at the end of two weeks and near castrate levels after 28 days. Patients randomized to enzalutamide (Arm B) will receive daily oral dose of 160 mg. Each cycle is defined as 28 days.

Patients will have Prostate-specific antigen level and symptoms assessment checked every cycle. Every 3 cycles patients will have repeat bone/CT scans to evaluate treatment response status. On CT scan, radiographic progression will be defined by RECIST criteria (i.e. >20% increase in the sum of target lesions). On bone scan, radiographic progression will be defined by PCWG2 criteria as ≥ 2 new bone lesions. However, for the first reassessment scan only, patients should remain on study and have a confirmatory scan performed 12 weeks (3 cycles) later. If this confirmatory scan shows 2 or more additional new lesions, this defines progression. The date of progression is the date of the first reassessment bone scan. If the confirmatory scan does not show any additional new lesions, patient remains on study. If progression is observed on subsequent bone scans, a confirmatory scan is not required; the date of this bone scan is the date of progression.

Patients with Prostate-specific antigen progression but with disease response or stable disease on imaging studies will remain on study until radiographic or other clinical progression criteria are met. Patients with radiographic disease progression will not receive continued BAT (arm A) or enzalutamide (arm B) and will be eligible for crossover to the opposite therapy. Patients on the BAT arm A can cross over to receive enzalutamide at time of progression or can choose to go off study and be treated with other standard of care treatments. Patients on the enzalutamide arm B will be allowed to cross-over to receive BAT or can choose to go off study and be treated with other standard of care treatments.

Patients with clinical progression due to prostate cancer must meet study exclusion criteria to be permitted to cross-over to the opposite treatment. Patients with clinical progression due to pain from prostate cancer are not permitted to cross-over.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group Performance status ≤2
* Age ≥18 years
* Histologically-confirmed adenocarcinoma of the prostate
* Treated with continuous androgen ablative therapy (either surgical castration or luteinizing hormone-releasing hormone agonist/antagonist)
* Documented castrate level of serum testosterone (<50 ng/dl)
* Metastatic disease radiographically documented by CT/MRI or bone scan.
* Must have had disease progression while on abiraterone acetate alone or abiraterone acetate in combination with other investigational agents based on:

  * Prostate-specific antigen progression defined as an increase in Prostate-specific antigen, as determined by 2 separate measurements taken at least 1 week apart

And/Or

* Radiographic disease progression, based on RECIST 1.1 in patients with measurable soft tissue lesions, or PCWG2 for patients with bone disease

  * Screening Prostate-specific antigen must be ≥ 1.0 ng/mL.
  * Prior treatment with additional second line hormone therapies is allowed.
  * No prior treatment with enzalutamide, Apalutamide (ARN-509), Darolutamide (ODM-201), galeterone or other investigational androgen receptor targeted treatment is allowed.
  * Prior docetaxel for hormone-sensitive prostate cancer is permitted if ≤ 6 doses were given in conjunction with first-line androgen deprivation therapy and >12 months since last dose of docetaxel.
  * Prior treatment with Provenge vaccine and 223Radium (Xofigo) is allowed if >4 weeks from last dose.
  * Patients must be withdrawn from abiraterone for ≥ 2 weeks.
  * Patients must be weaned off prednisone and be off therapy for ≥ 1 week prior to starting therapy.
  * Acceptable liver function:
* Bilirubin < 2.5 times institutional upper limit of normal (ULN)
* aspartate aminotransferase (SGOT) and alanine aminotransferase (SGPT) < 2.5 times ULN

  - Acceptable renal function:
* Serum creatinine < 2.5 times ULN

  - Acceptable hematologic status:
* Absolute neutrophil count (ANC) ≥ 1500 cells/mm3 (1.5 ×109/L)
* Platelet count ≥ 100,000 platelet/mm3 (100 ×109/L)
* Hemoglobin ≥ 9 g/dL.

  * At least 4 wks since prior radiation.
  * Ability to understand and willingness to sign a written informed consent document.
  * Patients on either treatment arm will be considered for crossover if they demonstrate evidence of radiographic disease progression.

Exclusion Criteria:

* Pain due to metastatic prostate cancer requiring treatment intervention.
* Eastern Cooperative Oncology Group Performance status ≥3
* Prior treatment with enzalutamide is prohibited
* Prior treatment with docetaxel or cabazitaxel for metastatic castration-resistant prostate cancer is prohibited.
* Requires urinary catheterization for voiding due to obstruction secondary to prostatic enlargement well documented to be due to prostate cancer or benign prostatic hyperplasia (BPH).
* Evidence of disease in sites or extent that, in the opinion of the investigator, would put the patient at risk from therapy with testosterone (e.g. femoral metastases with concern over fracture risk, severe and extensive spinal metastases with concern over spinal cord compression, extensive liver metastases)
* Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study
* Active uncontrolled infection, including known history of HIV/AIDS or hepatitis B or C.
* Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule.
* Patients receiving anticoagulation therapy with Coumadin are not eligible for study. [Patients on non-coumadin anticoagulants (Lovenox, Xarelto, etc.) are eligible for study. Patients on Coumadin who can be transitioned to lovenox prior to starting study treatments will be eligible].
* Patients with prior history of a thromboembolic event within the last 12 months that is not being treated with systemic anticoagulation are excluded.
* Patients allergic to sesame seed oil or cottonseed oil are excluded.
* Major surgery (eg, requiring general anesthesia) within 3 weeks before screening, or has not fully recovered from prior surgery (ie, unhealed wound). Note: subjects with planned surgical procedures to be conducted under local anesthesia may participate.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2015-01; Primary Completion 2018-10-26 (Actual); Study Completion 2020-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Denmeade, MD, Principal Investigator — Johns Hopkins School of Medicine - Sidney Kimmel Comprehensive Cancer Center
Locations (17):
- United States (17):
  - Unversity of Alabama, Birmingham, Alabama
  - City of Hope, Duarte, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Piedmont Cancer Institute, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Tulane University Medical Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - SKCCC at Johns Hopkins, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Neraska Cancer Specialists, Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Washing, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Denmeade SR, Wang H, Agarwal N, Smith DC, Schweizer MT, Stein MN, Assikis V, Twardowski PW, Flaig TW, Szmulewitz RZ, Holzbeierlein JM, Hauke RJ, Sonpavde G, Garcia JA, Hussain A, Sartor O, Mao S, Cao H, Fu W, Wang T, Abdallah R, Lim SJ, Bolejack V, Paller CJ, Carducci MA, Markowski MC, Eisenberger MA, Antonarakis ES. TRANSFORMER: A Randomized Phase II Study Comparing Bipolar Androgen Therapy Versus Enzalutamide in Asymptomatic Men With Castration-Resistant Metastatic Prostate Cancer. J Clin Oncol. 2021 Apr 20;39(12):1371-1382. doi: 10.1200/JCO.20.02759. Epub 2021 Feb 22. PMID 33617303

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 27 participants were not assigned to intervention due to screen failure, withdrawn consent, or PI decision.
Period: Overall Study
Arm/Group | Arm A: Testosterone Cypionate or Testosterone Enanthate | Arm B: Enzalutamide
Started | 94 | 101
Completed | 94 | 101
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Testosterone Cypionate or Testosterone Enanthate | Arm B: Enzalutamide | Total
Number analyzed (Participants) | 94 | 101 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (8.05) | 70.4 (7.59) | 70.5 (7.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 94 | 101 | 195
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 3 | 5
  Black or African American | 7 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 82 | 88 | 170
  Other | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 94 | 101 | 195
Weight (kg) [Mean (Standard Deviation); unit: Kilogram] | 93.8 (17.7) | 94.4 (19.7) | 94.1 (18.7)
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 176.5 (7.26) | 175.2 (12.4) | 175.8 (10.2)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilogram per meter square (Kg/m^2)] — Population: Data collected for BMI in 93/94 at Arm A and 95/101 at Arm B.
  Kilogram per meter square (Kg/m^2)
    number analyzed (Participants) | 93 | 95 | 188
    (all) | 29.9 (5.96) | 29.7 (7.17) | 29.8 (6.58)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG scale measures performance status, with scores ranging from 0-5; 0= fully active, performs without restriction, 1= can ambulate, but restricted in physically strenuous activity, 2= ambulatory and capable of self-care, but unable to work, active for >50% of waking hours, 3= limited self-care, confined to bed or chair for >50% of waking hours, 4= completely disabled, totally confined to bed/chair, 5= deceased Population: Data collected for ECOG performance status in 99/101 at Arm B.
  Participants
    0: number analyzed (Participants) | 94 | 99 | 193
    0 | 53 | 73 | 126
    1 | 40 | 25 | 65
    2 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival as Measured by Number of Months Until Clinical or Radiographic Progression
Description: Time to clinical progression will be defined as months from randomization to any of the following (whichever occurs earlier):
  * Cancer pain requiring initiation of chronic administration of opiate analgesia (oral opiate use for ≥3 weeks; parenteral opiate use for ≥7 days. Patients with cancer pain requiring opiate analgesia for relief should also be assessed by the investigator for the need for initiating systemic chemotherapy or palliative radiation.
  * Development of a skeletal-related event (SRE): pathologic fracture, spinal cord compression, or need for surgical intervention or radiation therapy to the bone.
  * Development of clinically significant symptoms due to loco-regional tumor progression (e.g. urinary obstruction) requiring surgical intervention or radiation therapy.
Time Frame: up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: Testosterone Cypionate or Testosterone Enanthate | Arm B: Enzalutamide
Number analyzed (Participants) | 94 | 101
months | 5.62 [4.76 to 5.91] | 5.72 [3.78 to 8.34]

2. Secondary Outcome: Radiographic Progression
Description: Number of months until 20% increase in the sum of target lesions on CT scans.
Time Frame: up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: Testosterone Cypionate or Testosterone Enanthate | Arm B: Enzalutamide
Number analyzed (Participants) | 94 | 101
months | 5.75 [5.55 to 8.41] | 8.28 [5.52 to 11.07]

3. Secondary Outcome: Prostate-Specific Antigen Response Rate
Description: Number of participants achieving a Prostate-Specific Antigen decline ≥ 50% according to Prostate Cancer Working Group (PCWG2) criteria.
Time Frame: Up to 2 years
Population: Data was not evaluable for this outcome measure in 7/94 participants from arm A and 7/101 participants from arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Testosterone Cypionate or Testosterone Enanthate | Arm B: Enzalutamide
Number analyzed (Participants) | 87 | 94
Participants | 14 | 18

4. Secondary Outcome: Objective Response Rate as Determined by RECIST
Description: Number of participants with partial (PR) or complete response (CR) as defined by response evaluation criteria in solid tumors (RECIST), where CR is a disappearance of all target lesions and PR is ≥30% reduction in the sum of the longest diameter of target lesions.
Time Frame: Up to 2 years
Population: Only participants with at least one post-baseline assessment were included to assess this outcome measure. Data was not evaluable in 61/94 participants from arm A and 77/101 participants from arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Testosterone Cypionate or Testosterone Enanthate | Arm B: Enzalutamide
Number analyzed (Participants) | 33 | 24
Participants | 8 | 1

5. Secondary Outcome: Time to Prostate-Specific Antigen Progression
Description: Reported as number of months till Prostate-Specific Antigen increase of greater or equal to 50% according to Prostate Cancer Working Group (PCWG2) criteria.
Time Frame: Up to 2 years
Population: Date is not evaluable for this outcome measure in 3/94 participants from arm A and 3/101 participants from arm B.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Arm A: Testosterone Cypionate or Testosterone Enanthate | Arm B: Enzalutamide
Number analyzed (Participants) | 91 | 98
month | 2.79 [1.81 to 4.50] | 3.81 [2.76 to 5.59]

6. Secondary Outcome: Quality of Life as Assessed by the Positive Affect Score of the Positive and Negative Affect Schedule (PANAS)
Description: The Positive Affect Score is calculated by adding the scores on items 1, 3, 5, 9, 10, 12, 14, 16, 17, and 19. Scores can range from 10 - 50, with higher scores representing higher levels of positive affect.
Time Frame: up to 1 year
Population: Questionnaires were not completed by all participants. Therefore, data was only collected from: Arm A- 87/94 at baseline, 81/94 at month 1, 71/94 at month 3, 54/94 at month 6 and 17/94 at month 12. Arm B- 93/101 at baseline, 86/101 at month 1, 75/101 at month 3, 55/101 at month 6 and 25/101 at month 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Testosterone Cypionate or Testosterone Enanthate | Arm B: Enzalutamide
Number analyzed (Participants) | 94 | 101
score on a scale
  Baseline: number analyzed (Participants) | 87 | 93
  Baseline | 33.99 (8.69) | 32.35 (8.58)
  Month 1: number analyzed (Participants) | 81 | 86
  Month 1 | 33.72 (8.46) | 32.33 (7.75)
  Month 3: number analyzed (Participants) | 71 | 75
  Month 3 | 33.23 (9.34) | 31.48 (7.67)
  Month 6: number analyzed (Participants) | 54 | 55
  Month 6 | 33.96 (9.80) | 31.84 (7.81)
  Month 12: number analyzed (Participants) | 17 | 25
  Month 12 | 36.24 (5.66) | 29.88 (8.54)

7. Secondary Outcome: Quality of Life as Assessed by the Negative Affect Score of the Positive and Negative Affect Schedule (PANAS)
Description: The Negative Affect Score is calculated by adding the scores on items 2, 4, 6, 7, 8, 11, 13, 15, 18, and 20. Scores can range from 10 - 50, with lower scores representing lower levels of negative affect.
Time Frame: up to 1 year
Population: Questionnaires were not completed by all participants. Therefore, data was only collected from: Arm A- 87/94 at baseline, 81/94 at month 1, 71/94 at month 3, 54/94 at month 6 and 17/94 at month 12.Arm B- 93/101 at baseline, 86/101 at month 1, 75/101 at month 3, 55/101 at month 6 and 25/101 at month 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Testosterone Cypionate or Testosterone Enanthate | Arm B: Enzalutamide
Number analyzed (Participants) | 94 | 101
score on a scale
  Baseline: number analyzed (Participants) | 87 | 93
  Baseline | 13.89 (4.89) | 13.96 (4.75)
  Month 1: number analyzed (Participants) | 81 | 86
  Month 1 | 14.28 (5.81) | 14.90 (6.16)
  Month 3: number analyzed (Participants) | 71 | 75
  Month 3 | 14.44 (5.52) | 15.43 (6.54)
  Month 6: number analyzed (Participants) | 54 | 55
  Month 6 | 14.26 (6.13) | 14.80 (6.20)
  Month 12: number analyzed (Participants) | 17 | 25
  Month 12 | 14.24 (6.45) | 13.48 (3.64)

8. Secondary Outcome: Change in Quality of Life as Assessed by the International Index of Erectile Function (IIEF) Questionnaire
Description: The IIEF assesses erectile function (EF), orgasmic function (OF), sexual desire (SD), intercourse satisfaction (IS), orgasmic satisfaction (OS). Each of domains are scored on a scale of 0 to 5 with a lower score indicating a bad quality sex life. The IIEF questionnaire has a total score that ranges from 5 to 25 with lower score indicating less erectile dysfunction. A positive change in the score reflects better outcome.
Time Frame: up to 1 year
Population: Questionnaires were not completed by all participants. Therefore, data was only collected from: Arm A- 72/94 at baseline to month 1, 63/94 at month 3, 42/94 at month 6, and 14/94 at month 12. Arm B- 74/101 at month 1, 57/101 at month 3, 46/101 at month 6 and 20/101 at month 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Testosterone Cypionate or Testosterone Enanthate | Arm B: Enzalutamide
Number analyzed (Participants) | 94 | 101
score on a scale
  EF - baseline to month 1: number analyzed (Participants) | 72 | 74
  EF - baseline to month 1 | 1.17 (4.56) | 0.09 (1.84)
  EF - baseline to month 3: number analyzed (Participants) | 63 | 57
  EF - baseline to month 3 | 2.65 (6.46) | 0.05 (2.86)
  EF - baseline to month 6: number analyzed (Participants) | 42 | 46
  EF - baseline to month 6 | 2.36 (6.30) | 0.65 (3.75)
  EF - baseline to month 12: number analyzed (Participants) | 14 | 20
  EF - baseline to month 12 | 2.5 (6.95) | 0.05 (1.32)
  OF - baseline to month 1: number analyzed (Participants) | 74 | 80
  OF - baseline to month 1 | 0.91 (2.39) | 0.25 (1.13)
  OF - baseline to month 3: number analyzed (Participants) | 67 | 65
  OF - baseline to month 3 | 1.93 (2.99) | -0.02 (1.22)
  OF - baseline to month 6: number analyzed (Participants) | 47 | 53
  OF - baseline to month 6 | 2.19 (3.48) | 0.04 (1.21)
  OF - baseline to month 12: number analyzed (Participants) | 15 | 24
  OF - baseline to month 12 | 2.93 (3.86) | 0.17 (0.82)
  SD - baseline to month 1: number analyzed (Participants) | 75 | 74
  SD - baseline to month 1 | 0.97 (2.09) | -0.27 (1.55)
  SD - baseline to month 3: number analyzed (Participants) | 66 | 61
  SD - baseline to month 3 | 1.85 (2.70) | 0.10 (1.51)
  SD - baseline to month 6: number analyzed (Participants) | 46 | 51
  SD - baseline to month 6 | 2.52 (2.59) | 0.18 (1.77)
  SD - baseline to month 12: number analyzed (Participants) | 16 | 20
  SD - baseline to month 12 | 2.38 (2.31) | 0.30 (1.49)
  IS - baseline to month 1: number analyzed (Participants) | 76 | 78
  IS - baseline to month 1 | 0.36 (2.60) | -0.01 (1.59)
  IS - baseline to month 3: number analyzed (Participants) | 69 | 65
  IS - baseline to month 3 | 1.55 (4.83) | 0.05 (1.66)
  IS - baseline to month 6: number analyzed (Participants) | 47 | 51
  IS - baseline to month 6 | 0.74 (4.18) | 0.08 (1.94)
  IS - baseline to month 12: number analyzed (Participants) | 15 | 23
  IS - baseline to month 12 | 2.40 (4.73) | 0.00 (0.00)
  OS - baseline to month 1: number analyzed (Participants) | 68 | 72
  OS - baseline to month 1 | 0.65 (2.23) | 0.17 (1.94)
  OS - baseline to month 3: number analyzed (Participants) | 60 | 55
  OS - baseline to month 3 | 1.13 (2.70) | 0.25 (1.71)
  OS - baseline to month 6: number analyzed (Participants) | 42 | 46
  OS - baseline to month 6 | 0.60 (3.09) | -0.09 (1.50)
  OS - baseline to month 12: number analyzed (Participants) | 12 | 20
  OS - baseline to month 12 | 2.00 (3.67) | 0.20 (1.47)

9. Secondary Outcome: Quality of Life as Assessed by Short Form 36
Description: All questions are scored on a scale from 0 to 100. The total score from all of the questions answered is divided by the total number of the questions answered yielding a global score from 0-100 with 100 representing the highest level of functioning possible.
Time Frame: up to 1 year
Population: Questionnaires were not completed by all participants. Therefore, data was only collected from: Arm A- 89/94 at baseline, 84/94 at month 1, 74/94 at month 3, 55/94 at month 6 and 18/94 at month 12.Arm B- 96/101 at baseline, 86/101 at month 1, 81/101 at month 3, 56/101 at month 6 and 25/101 at month 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Testosterone Cypionate or Testosterone Enanthate | Arm B: Enzalutamide
Number analyzed (Participants) | 94 | 101
score on a scale
  Baseline: number analyzed (Participants) | 89 | 96
  Baseline | 63.16 (12.7) | 61.89 (11.9)
  Month 1: number analyzed (Participants) | 84 | 86
  Month 1 | 61.68 (11.7) | 56.94 (13.6)
  Month 3: number analyzed (Participants) | 74 | 81
  Month 3 | 62.34 (13.8) | 55.34 (15.1)
  Month 6: number analyzed (Participants) | 55 | 56
  Month 6 | 63.49 (13.3) | 58.67 (13.6)
  Month 12: number analyzed (Participants) | 18 | 25
  Month 12 | 67.35 (9.45) | 59.65 (14.9)

10. Secondary Outcome: Quality of Life as Assessed by FACIT Fatigue Scale
Description: The Functional Assessment of Chronic Illness Therapy - Fatigue has a score range of 0-52 with higher scores indicating better quality of life.
Time Frame: up to 1 year
Population: Questionnaires were not completed by all participants. Therefore, data was only collected from: 84/94 at month 1, 76/94 at month 3, 55/94 at month 6 and 18/94 at month 12.Arm B- 87/101 at month 1, 81/101 at month 3, 56/101 at month 6 and 25/101 at month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Testosterone Cypionate or Testosterone Enanthate | Arm B: Enzalutamide
Number analyzed (Participants) | 94 | 101
score on a scale
  Month 1: number analyzed (Participants) | 84 | 87
  Month 1 | 38.13 (9.85) | 32.60 (12.0)
  Month 3: number analyzed (Participants) | 76 | 81
  Month 3 | 38.39 (11.1) | 33.51 (11.8)
  Month 6: number analyzed (Participants) | 55 | 56
  Month 6 | 39.23 (11.4) | 34.51 (11.3)
  Month 12: number analyzed (Participants) | 18 | 25
  Month 12 | 41.67 (8.39) | 34.58 (13.5)

11. Secondary Outcome: Pain Severity as Assessed by the Brief Pain Inventory
Description: Severity is calculated by adding the scores for questions 2, 3, 4 and 5 and then dividing by 4. This gives a severity score out of 10, high score indicates more severe pain.
Time Frame: 1 year
Population: For Arm A, the data was only collected from 85/94 at baseline, 78/94 at month 1, 67/94 at month 3, 54/94 at month 6, 17/94 at month 12.
  For Arm B, the data was only collected from 92/101 at baseline, 82/101 at month 1, 76/101 at month 3, 54/101 at month 6, 24/101 at month 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Testosterone Cypionate or Testosterone Enanthate | Arm B: Enzalutamide
Number analyzed (Participants) | 94 | 101
score on a scale
  Baseline: number analyzed (Participants) | 85 | 92
  Baseline | 1.29 (1.99) | 1.20 (1.92)
  Month 1: number analyzed (Participants) | 78 | 82
  Month 1 | 1.19 (1.85) | 1.94 (2.19)
  Month 3: number analyzed (Participants) | 67 | 76
  Month 3 | 1.67 (2.06) | 1.62 (2.05)
  Month 6: number analyzed (Participants) | 54 | 54
  Month 6 | 1.57 (2.12) | 1.81 (2.18)
  Month 12: number analyzed (Participants) | 17 | 24
  Month 12 | 0.76 (1.39) | 1.13 (1.87)

12. Secondary Outcome: Pain Interference as Assessed by the Brief Pain Inventory
Description: Interference is calculated by adding the scores for questions 8a, b, c, d, e, f and g and then dividing by 7. This gives an interference score out of 10, higher score indicates more pain interference.
Time Frame: 1 year
Population: For Arm A, the data was only collected from 82/94 at baseline, 78/94 at month 1, 65/94 at month 3, 53/94 at month 6, 17/94 at month 12.
  For Arm B, the data was only collected from 91/101 at baseline, 81/101 at month 1, 76/101 at month 3, 55/101 at month 6, 25/101 at month 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Testosterone Cypionate or Testosterone Enanthate | Arm B: Enzalutamide
Number analyzed (Participants) | 94 | 101
score on a scale
  Baseline: number analyzed (Participants) | 82 | 91
  Baseline | 1.22 (1.77) | 1.27 (1.87)
  Month 1: number analyzed (Participants) | 78 | 81
  Month 1 | 1.55 (2.00) | 2.26 (2.52)
  Month 3: number analyzed (Participants) | 65 | 76
  Month 3 | 2.00 (2.20) | 1.94 (2.26)
  Month 6: number analyzed (Participants) | 53 | 55
  Month 6 | 1.96 (2.59) | 1.84 (2.07)
  Month 12: number analyzed (Participants) | 17 | 25
  Month 12 | 1.04 (1.85) | 1.70 (2.39)

13. Secondary Outcome: Overall Survival
Description: Time until death for any reasons
Time Frame: up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Testosterone Cypionate or Testosterone Enanthate | Arm B: Enzalutamide
Number analyzed (Participants) | 94 | 101
months | 32.9 [28.2 to 37.3] | 29 [26.2 to 35.5]

14. Secondary Outcome: Progression Free Survival on Crossover Treatment
Description: Time from initiation of therapy to progression on crossover treatment
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Testosterone Cypionate or Testosterone Enanthate | Arm B: Enzalutamide
Number analyzed (Participants) | 94 | 101
months | 28.2 [23.6 to NA] — Not reached | 19.6 [12.9 to 29.7]

ADVERSE EVENTS:
Time Frame: up to 2 years
Arm/Group | Arm A: Testosterone Cypionate or Testosterone Enanthate | Arm B: Enzalutamide
All-Cause Mortality (participants affected / at risk) | 0/94 | 1/101
Serious Adverse Events (participants affected / at risk) | 4/94 | 11/101
Other Adverse Events (participants affected / at risk) | 22/94 | 29/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Testosterone Cypionate or Testosterone Enanthate (N=94) | Arm B: Enzalutamide (N=101)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
myocardial infarction (Cardiac disorders) | 0 (0) | 1 (2) — ST elevation myocardial infarction (cardiac cauterization with stent placement)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Testosterone Cypionate or Testosterone Enanthate (N=94) | Arm B: Enzalutamide (N=101)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 6 (6)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 3 (3) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8)
fatigue (General disorders) | 11 (11) | 3 (3)
pain (General disorders) | 4 (4) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT02286921/SAP_001.pdf
  • Study Protocol (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT02286921/Prot_002.pdf